CLINICAL TRIAL: NCT06698081
Title: The Effect of Using Multimedia During the Informed Consent Process on the Anxiety of Parents of Orchiopexy Patients: a Randomized Controlled Trial
Brief Title: The Effect of Using Multimedia During the Informed Consent Process on the Anxiety of Parents of Orchiopexy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MAR.UAD.009
Record Dates: First submitted 2024-11-12; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Undescended Testis; Anxiety State
Keywords: undescended testis; anxiety state
MeSH Terms: conditions — Cryptorchidism; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Informed Consent Form + Verbal Information (No Intervention): The first group will be informed of the Standard Informed Consent Form and Verbal Information during the preoperative process.
- Standard Informed Consent Form + Verbal Information + Multimedia (Active Comparator): The second group will be informed of the Standard Informed Consent Form, Verbal Information, and Multimedia.
  Interventions: Other: Video Multimedia

INTERVENTIONS:
Other: Video Multimedia — The second group will be informed of the Standard Informed Consent Form, Verbal Information, and Multimedia. In addition to the standard consent process, we planned to show a 6-minute video multimedia presentation containing information about undescended testis and orchiopexy.
  Other Names: Multimedia Group
  Arms: Standard Informed Consent Form + Verbal Information + Multimedia

SUMMARY:
Aim: The goal of this randomized controlled trial is to detect the effect of using multimedia during the informed consent process on the anxiety of parents of orchiopexy patients.

Parents (primary caregivers) of the patients who underwent orchiopexy surgery are included in the study.

The main question it aims to answer is:

• Does the use of multimedia during the preoperative consent process affect the anxiety level of parents of patients undergoing orchiopexy surgery?

DETAILED DESCRIPTION:
Aim: The goal of this randomized controlled trial is to detect the effect of using multimedia during the informed consent process on the anxiety of parents of orchiopexy patients.

Parents (primary caregivers) of the patients who underwent orchiopexy surgery are included in the study.

The patient's age, gender, known diseases, previous hospital admissions, and whether they have undergone surgery before will be recorded. The primary caregiver's age, gender, known diseases, educational status, occupation, number of children, and any additional illnesses in other children will be noted.

Patients will be randomized into 2 groups with the help of (https://www.randomizer.org/ ). The first group will be informed of the Standard Consent Form and Verbal Information during the preoperative process. In contrast, the second group will be informed of the Standard Consent Form, Verbal Information, and Multimedia. Both groups will fill out the Hospital Anxiety and Depression Scale(HADS), BECK Anxiety Inventory(BAI), and The State-Trait Anxiety Inventory (STAI) Form Tx 1-2 forms one day before the surgery and on the 7th day after the surgery to determine their anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* parents of orchiopexy patients

Exclusion Criteria:

* history of previous orchiopexy surgery
* orchiopexy with other surgical procedures ( f.e. Hypospadias repair)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-03-25 (Estimated); Study Completion 2025-03-28 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 1 week
  The participants' HADS scores will be noted one day before the surgery and on the 7th day after the surgery.
Beck Anxiety Inventory | 1 week
  The participants' BECK anxiety scores will be noted one day before the surgery and on the 7th day after the surgery.
State-Trait Anxiety Inventory (STAI) | 1 week
  The participants' STAI - Tx I and STAI -Tx II scores will be noted one day before and on the 7th day after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Cagri Akin Sekerci, Study Director — Marmara University
Locations (1):
- Marmara University School of Medicine, Department of Urology, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No